CLINICAL TRIAL: NCT06041594
Title: Treating Pulmonary Embolism With Laguna Thrombectomy System (TRUST)
Acronym: TRUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innova Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001 Rev. C
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Embolism
Keywords: Laguna Thrombectomy System; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laguna Thrombectomy System (Experimental)
  Interventions: Device: Laguna Thrombectomy System

INTERVENTIONS:
Device: Laguna Thrombectomy System — Removal of clot using the Laguna Thrombectomy System to treat Pulmonary Embolism

SUMMARY:
This is a prospective, multi-center, pivotal study to demonstrate the safety and effectiveness of the Laguna Thrombectomy System for the treatment of pulmonary embolism. The Laguna Thrombectomy System is an investigational device which consists of the Laguna Clot Retriever™ System and the Malibu Aspiration Catheter™ System. These devices are manufactured by Innova Vascular, Inc.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age; < 85 years old
2. RV/LV ratio > 0.9 as determined by CTA
3. Systolic blood pressure > 90 mmHg
4. Heart rate ≤ 120
5. Patient is deemed eligible for procedure by the interventional investigator
6. CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery)
7. PE Symptom duration ≤ 14 days

Exclusion Criteria:

1. Systolic pulmonary artery pressure > 70 mmHg on initial invasive hemodynamic assessments
2. Life expectancy of < 90 days in the opinion of investigator at the time of enrollment
3. Subject pregnant or breast feeding
4. Current participation in another drug or medical device treatment study
5. In active chemotherapy or radiation treatment for a malignancy during the course of the study
6. Any intravascular administration of a fibrinolytic agent (such as Alteplase or Tenecteplase) within the last 30 days
7. Presence of recently placed (<8 weeks) intracardiac devices (such as pacemaker leads) in the right ventricle or right atrium
8. History of prior PE within the past 90 days
9. FiO2 Requirement: > 40% (6 LPM) to keep oxygen saturation > 90%
10. Hematocrit: < 28%
11. Platelets: < 100,000/microliter
12. Serum Creatinine: > 2 mg/dL
13. International Normalized Ratio (INR): > 3
14. Major Trauma Injury Severity Score (ISS): > 15
15. Cardiovascular or pulmonary surgery within the last 7 days
16. Known bleeding diathesis or coagulation disorder that cannot be managed with anti-coagulation
17. History of known severe or chronic pulmonary arterial hypertension
18. History or chronic left heart disease with left ventricular ejection fraction < 30%
19. History of underlying lung disease that is oxygen dependent
20. History of chest irradiation
21. Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
22. Any absolute contraindication to systemic or therapeutic dosage of heparin or anticoagulants
23. Imaging or other evidence that suggests, in the opinion of the investigator, the subject is not appropriate for mechanical thrombectomy intervention (e.g., inability to navigate to target location, predominantly chronic clot or non-clot embolus)
24. Known presence of clot in transit within right atrium or ventricle

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
A composite of the following major adverse events occurring within 48 (± 8) hours post-procedure: | within 48 (± 8) hours post-procedure
  * Device-related death within 48 (± 8) hours post-procedure
  * Major bleeding as defined by GUSTO (moderate or severe) within 48 (± 8) hours post-procedure.
  * The following treatment-related adverse events within 48 (± 8) hours post-procedure:
    * Cardio-respiratory deterioration,
    * Pulmonary vascular injury, and/or
    * Cardiac injury
Reduction in RV/LV ratio from baseline to 48 (± 8) hours (or at discharge, whichever occurs first) as assessed by Computed Tomography Angiography (CTA) | from baseline to 48 (± 8) hours (or at discharge, whichever occurs first)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (10):
  - University of California Irvine, Irvine, California
  - Memorial Care Long Beach Medical Center, Long Beach, California
  - Mission Hospital Regional Medical Center, Mission Viejo, California
  - St. Joseph Hospital of Orange, Orange, California
  - George Washington University, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Albany Medical Center, Albany, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Turkey (Türkiye) (4):
  - Ankara Bilkent City Hospital, Ankara
  - Hacettepe University Hospital, Ankara
  - Sancaktepe Sehit Prof. Dr. Ilhan Varan Training and Research Hospital, Istanbul
  - Dokuz Eylul University Research and Application Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No